CLINICAL TRIAL: NCT05779748
Title: The Effect of an Acute Bout of Exercise on Pain Sensitivity and Clinical Pain in Adults With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taif University (Other)
Collaborators: King Abdullah Hospital (Unknown)
Responsible Party: Principal Investigator, Hosam Alzahrani, Assistant Professor, Taif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIS-23-00007-11012023
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2023-03

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Isometric exercise-one repetition (Experimental): Isometric exercise consisting of 1 session only. The session will last for around 5 minutes which will include asking the patient to do 1 repetition of wall squat for 3 min or to volitional fatigue at 100° knee angle.
  Intervention: Other: Single bout of exercise
  Interventions: Other: Single bout of exercise
- Isometric exercise-three repetitions (Experimental): isometric exercise consisting of 1 session only. The session will last for around 10 minutes which will include asking the patient to perform 3 repetitions of wall squats (each time the exercise will be performed for 3 min or to volitional fatigue at 100°degree knee angle); the patient will be given 30-sec rest between repetitions.
  Intervention: Other: Single bout of exercise
  Interventions: Other: Single bout of exercise
- Control (No Intervention): Will not receive any intervention

INTERVENTIONS:
Other: Single bout of exercise — isometric wall squat at a knee joint angle of 100 degrees. Instruct participant to place their back against the wall with feet positioned parallel and spaced shoulder-width apart. Lower themselves down until they reached a knee joint angle of 100 degrees. Measure knee joint angle by placing a goniometer on the lateral epicondyle of the knee, in line with the femur whilst the anchor arm was in line with the lateral malleolus.
  Arms: Isometric exercise-one repetition; Isometric exercise-three repetitions

SUMMARY:
The goal of this interventional study is to investigate the efficacy of an acute bout of exercises on pain sensitivity (primary aim) and clinical pain intensity (secondary aim) among adults with Chronic Low Back Pain. The following question will be answered in this research Q1: Is acute bout of exercise effective in reducing pain among adults with Chronic Low Back Pain?

Participants who agree to participate and sign the informed consent will be randomized to one of three groups:

Group 1: Isometric exercise with neutral language and no verbal suggestion consisting of 1 rep of wall squat, 3 min or to volitional fatigue at 100° knee angle;(n=30).

Group 2: Isometric exercise with neutral language and no verbal suggestion consisting of 3 reps of wall squat, 3 min or to volitional fatigue at 100°degree knee angle, 30-sec rest between rep, ;(n=30).

Group 3 (Control group): true control (do nothing);(n=30).

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years or older; and
2. diagnosed with chronic non-specific LBP (lasting for more than 12 weeks).
3. Able to perform physical therapy exercises.

Exclusion Criteria:

1. pregnancy.
2. patients who have neurological compromise (e.g., cauda equine syndrome or spinal nerve compromise).
3. Patients who have spinal pathologies (e.g., fracture, ankylosing spondylitis)
4. Uncontrolled diabetic.
5. who has any history of heart disease (e.g., myocardial infarction, embolism)
6. Orthopaedic impairment (e.g., balance problems)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 Years to 65 Years (Adult, Older Adult)
Enrollment: 90 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-08-05 (Actual)

PRIMARY OUTCOMES:
Pain pressure threshold | [ Time Frame: Change from pre-intervention (baseline) compared to post-intervention (immediately after session) ]
  The pain will be measured using digital pressure algometer, FDX®️ (Wagner instrument, Greenwich, USA). All trials will be conducted on forearm, lumbar spine and calf sites. There will be at least 20 sec rest before an individual site is tested again. Two trials will be performed at each site. The raw values of each test will be recorded.
  Because we are testing repeated times, we will use a marker to mark the location of each test site to ensure consistency in location.
  Algometer must be positioned perpendicular to the measurement site for all trials.

SECONDARY OUTCOMES:
Pain intensity | [ Time Frame: Change from pre-intervention (baseline) compared to post-intervention (immediately after session) ]
  It will be assessed using Visual Analogue Scale (VAS; 0-10). A rating of zero means that participant don't currently have pain at the low back. A rating of ten on this scale means that the pain at low back is the worst pain. So, the higher the number on this scale means the higher the pain intensity participant is experiencing.

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Alzahrani, PhD, Principal Investigator — Taif University
Locations (1):
- King Abdullah Hospital, Bisha, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No